CLINICAL TRIAL: NCT06798272
Title: Measurement of Skinfold Thickness in Subscapular Area to Monitor Hydration Status in Chronic Hemodialysis Patients
Brief Title: Monitoring of Hydration Status in Chronic Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Michal Nowicki, Professor MD, Medical University of Lodz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 163/20
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis; Kidney Failure; Overhydration
Keywords: hemodialysis; water-electrolyte balance; dry body mass; skinfold thickness
MeSH Terms: conditions — Renal Insufficiency; Water Intoxication | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- changes of overhydration during hemodialysis session (Experimental)
  Interventions: Procedure: dialysisis with and without glucose in the dialysis

INTERVENTIONS:
Procedure: dialysisis with and without glucose in the dialysis — there were assessed three consecutive hemodialysis sessions

SUMMARY:
Background Maintaining fluid balance is one of major challenges of the dialysis therapy. It includes, in particular, the management of "dry body mass". We postulated that simple measurement of subscapular skinfold thickness before and after hemodialysis could help monitor hydration status in chronic dialysis patients.

Aim of the study The aim of the study was to compare the conventional methods of monitoring hydration status during hemodialysis with an assessment of skin fold thickness.

Materials and Methods 50 participants (21 F, 29 M; age 60 ±15 years) were enrolled. Directly before the hemodialysis session the following parameters were measured: body composition with bioimpedance spectroscopy, skinfold thickness in subscapular area with standardized caliper and blood tests: blood count, urea, n-terminal pro B-type natriuretic peptide (nt-proBNP) and pro-adrenomedullin (pro-ADM). The procedures were repeated at the end of three consecutive hemodialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis for at least 3 months

Exclusion Criteria:

* severe mental disabilities, poor compliance, any acute infection, instability of the cardiovascular hemodynamic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
changes in overhydration | From enrollment to one week

CONTACTS AND LOCATIONS:
Locations (1):
- Central University Hospital, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided